CLINICAL TRIAL: NCT02849938
Title: Evaluating the Value of Telehealth for Care of Children With Medical Complexity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CCCMCTeleMed
Record Dates: First submitted 2016-07-27; First posted 2016-07-29 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2017-04

CONDITIONS: Cerebral Palsy
Keywords: children with medical complexity; Telemedicine; Tracheostomy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (No Intervention): Usual care
- Telemedicine Group (Experimental): TytoCare Device
  Interventions: Device: TytoCare Device

INTERVENTIONS:
Device: TytoCare Device — Tyto is a handheld, mobile device designed for capture and transmission of ear/throat/skin images and lung/heart auscultations. It may be used to perform non-invasive, medical examinations, either on a patient (by another person, most commonly a family member, or by a medical professional) or self-performed by the patient, for remote review by a medical practitioner. It is suitable for use on patients in both clinical and home environment.
  Arms: Telemedicine Group

SUMMARY:
The specific aims of the study are to:

1. Assess the feasibility of a TytoCare telehealth device with remote audio/video connection for evaluation of children with medical complexity in the home environment.
2. Evaluate the usability of a TytoCare telehealth device in transmitting real time images (otoscope, oropharyngeal exam, camera), temperature, and sound (stethoscope for heart and breath sounds)
3. Compare the impact of the TytoCare telehealth device versus traditional telephone assessment on patient management and user satisfaction

DETAILED DESCRIPTION:
Eligible children of interested parent(s) will be randomly assigned to either the control group (standard care) or the intervention group (Tyto device). Randomization will be performed using an online randomization program to generate group assignments for the 25 subjects. Subjects will be stratified by whether they have a tracheostomy or not and be assigned 1.5:1 to achieve 15 children in the device group and 10 children in the control group. Informed consent will be obtained for children in each group.

Children/families in the control group will continue to get usual care through the CCCMC program, and will be able to access their providers via telephone for urgent care needs and scheduled follow up. For evaluation purposes, data collection will include the monthly encounter tracking that is done routinely as part of the CCCMC program, and research surveys completed by both parents and HCPs. Parents will complete a Parent Survey by phone once each month for the 3-month study period. The CCCMC HCPs will complete the Provider Survey electronic survey with each telephone encounter where the HCP would have liked to use the device.

For those assigned to the device group, parents will be instructed to contact their CCCMC HCP as usual, see bullet points above, when health concerns arise and their HCP will decide if she would like a telehealth visit. Telehealth/video visits may also be scheduled in advance as a matter of routine follow-up care. In the event that an exam is deemed necessary by the HCP, the parent or caregiver will be directed to connect via the remote exam device. The provider will conduct a 2-way live interactive audio/video visit with the patient. The parent or caregiver will use the remote exam device to provide temperature, lung sounds, heart sounds, oropharyngeal exam, skin exam and/or ear exam as clinically indicated. Direction for necessary treatment, referral to an ED, clinic or inpatient care will be at the discretion of the CCCMC provider. For evaluation purposes, in addition to the monthly encounter tracking that is done as part of the CCCMC program, both parents and HCPs will complete surveys. Parents will complete a Parent Survey by phone once each month for the 3-month study period. The CCCMC HCPs will complete the Provider Survey via a Qualtrics link with each telehealth encounter.

Additional data collected will include subject demographics, and encounter data that is routinely collected as a part of the CCCMC program. Images of patient encounters will be transmitted in real time via the telemedicine device encrypted software. Provider Survey data will be gathered via Qualtrics. Tyto will retain / store data obtained from device group encounters in a de-identified way for development purposes only.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 1 month to 18 years
* Patient currently enrolled in CCCMC program at ACH-OL
* Parental permission/consent
* English-speaking (at least one parent)
* Internet connected home wi-fi

Exclusion Criteria

* Unable to comply with study requirements

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2016-09; Primary Completion 2017-01-31 (Actual); Study Completion 2017-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia M Notario, MD, Principal Investigator — Advocate Children's Hospital

IPD SHARING:
Plan to Share IPD: No
Will share only aggregate and overall project results through poster and/or oral presentations at local, regional and national meetings.

REFERENCES:
- [Derived] Notario PM, Gentile E, Amidon M, Angst D, Lefaiver C, Webster K. Home-Based Telemedicine for Children with Medical Complexity. Telemed J E Health. 2019 Nov;25(11):1123-1132. doi: 10.1089/tmj.2018.0186. Epub 2019 Jan 30. PMID 30628860

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Received usual care through the pediatric complex care program at our institution. This included 24/7 availability by the program clinicians for phone calls and electronic message from caregivers. The clinicians provided primary care and consultative services focusing on outpatient comprehensive care visits. The team also provided inpatient consultation.
- Telemedicine Group: Received the TytoCare Device in addition to usual care.
  TytoCare Device: Tyto is a handheld, mobile device designed for capture and transmission of ear/throat/skin images and lung/heart auscultations. It may be used to perform non-invasive, medical examinations, either on a patient (by another person, most commonly a family member, or by a medical professional) or self-performed by the patient, for remote review by a medical practitioner. It is suitable for use on patients in both clinical and home environment.
Period: Overall Study
Arm/Group | Control Group | Telemedicine Group
Started | 9 | 15
Completed | 9 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Telemedicine Group | Total
Number analyzed (Participants) | 9 | 15 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 15 | 24
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.32 (6.67) | 8.81 (5.74) | 9.01 (6.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 3 | 8 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-white | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 9 | 15 | 24
Number of specialists involved in the care of the patient [Mean (Standard Deviation); unit: specialists] | 5.55 (1.87) | 5.87 (1.51) | 5.67 (1.69)
Trach: present [Count of Participants; unit: Participants] | 4 | 7 | 11
Number of medical diagnoses active at enrollment [Mean (Standard Deviation); unit: diagnoses] | 11 (3.71) | 10 (3.40) | 10 (3.57)

OUTCOME MEASURES:

1. Primary Outcome: Frequency of In-person Health Care Encounters
Description: Hospital day length of stay reported as the total number of hospital days in the group.
Time Frame: 3 months
Measure: Number; unit: days
Arm/Group | Control Group | Telemedicine Group
Number analyzed (Participants) | 9 | 15
days
  Hospitalization days - floor | 24 | 19
  Hospitalization days - ICU | 41 | 46

2. Secondary Outcome: Provider Survey
Description: Success of connection for telemedicine visits.
Time Frame: 3 months
Population: Control group participants did not have data for telemedicine device use as they did not have access to this.
Measure: Count of Units; unit: Visit Connections
Units Other Than Participants: Visit Connections
Arm/Group | Control Group | Telemedicine Group
Number analyzed (Participants) | 9 | 15
Number analyzed (Visit Connections) | 0 | 50
Visit Connections
  Connection worked great for telemedicine visit: number analyzed (Participants) | 0 | 15
  Connection worked great for telemedicine visit |  | 37
  Connection was problematic for telemedicine visit: number analyzed (Participants) | 0 | 15
  Connection was problematic for telemedicine visit |  | 9
  Not able to get connection with telemedicine visit: number analyzed (Participants) | 0 | 15
  Not able to get connection with telemedicine visit |  | 4

3. Secondary Outcome: Parent Survey
Description: Overall satisfaction with device, comfort with Device, satisfaction with clinician interactions and development of plans of care; Questions asked using 4 point Likert scale (4 = Very Satisfied , 1=Very Dissatisfied). Higher score more satisfaction
Time Frame: 3 months
Population: Control group participants did not answer questions regarding the tele health device in the satisfaction survey as they did not have access to this.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Control Group | Telemedicine Group
Number analyzed (Participants) | 9 | 15
units on a scale
  Satisfaction with telehealth device: number analyzed (Participants) | 0 | 15
  Satisfaction with telehealth device |  | 4 [3.5 to 4]
  Comfortable with telehealth device: number analyzed (Participants) | 0 | 15
  Comfortable with telehealth device |  | 4 [3.5 to 4]
  Interaction with clinicians | 4 [3.7 to 4] | 4 [4 to 4]
  Complex care program satisfaction | 4 [3.7 to 4] | 4 [4 to 4]

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Control Group | Telemedicine Group
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/15
Other Adverse Events (participants affected / at risk) | 0/9 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-29): https://cdn.clinicaltrials.gov/large-docs/38/NCT02849938/Prot_SAP_000.pdf